CLINICAL TRIAL: NCT02758236
Title: Tuberculosis Research of INA-RESPOND On Drug Resistance
Acronym: TRIPOD
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: INA102; U1111-1263-2311 (Other: WHO UTN Number)
Record Dates: First submitted 2016-04-04; First posted 2016-05-02 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Lung Tuberculosis; MDR TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects must be willing to allow storage of sputum, Mtb isolate, whole blood (PAXgene blood , plasma, PBMC), and urine on baseline, month 1, month 2, and end of treatment visit, saliva on baseline and end of treatment visit for use in future studies (for example, host response, spoligotyping, and genetic tests). Serum and whole blood for DNA are collected on baseline visit only.
  All samples will be stored at the NIHRD, Mtb isolate, plasma, saliva and urine will also be stored at each site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This study is a prospective observational cohort study of TB patients who are treated or evaluated at 10 study sites. Patients presenting with cough for 2 weeks or longer with at least one additional TB symptom and a chest X-ray suggestive of TB, will be invited to be enrolled in the study. The signed informed consent will designate their willingness to participate on this study.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study of TB patients who are treated or evaluated at 10 study sites. Patients presenting with cough for 2 weeks or longer with at least one additional TB symptom and a chest X-ray suggestive of TB, will be invited to be enrolled in the study. The signed informed consent will designate their willingness to participate on this study. Enrolled subjects will produce the sputum for bacteriological examination of M. tuberculosis by AFB, culture and Xpert. The sputum will also be tested by Xpert for drug resistance test. If the culture is positive, conventional DST will be performed, and M. tuberculosis isolates will be stored for spoligotyping and for future research on TB. All bacteriologicaly confirmed subjects will be followed for outcome assessment.

For all enrolled subjects chest X-ray results, demographic data, TB co-morbidities, symptoms, nutritional status, treatment regimens, compliance and outcome will be collected. In addition, sputum, blood and urine will also be collected for storage.

To estimate the proportion of MDR-TB amongst new and previously treated TB cases.

1. To evaluate accuracy of clinical diagnosis by comparing clinically defined TB to laboratory confirmed TB.
2. To compare AFB and Xpert MTB/RIF as TB diagnostic tests against culture result.
3. To estimate the sensitivity and specificity of Xpert MTB/RIF in detecting Rif susceptibility against DST.
4. To estimate the proportion of cured, completed, failed, died and lost to follow up as treatment outcomes on DS-TB and DR-TB cases
5. To evaluate the association of treatment success (cured or completed) with the following data:

   1. Demographics (age, sex)
   2. TB contact history
   3. Smoking habit
   4. Treatment seeking behavior
   5. Co-morbidities (HIV, DM)
   6. Primary and secondary drug resistance
   7. Symptoms
   8. Cavitary disease
   9. Nutritional status
   10. Treatment regimens
   11. Patient reported compliance
   12. Numbers of bacteria by AFB test
   13. TB strains (e.g Beijing)

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of having pulmonary TB
* Cough ≥ 2 weeks
* At least one other TB clinical symptom

  * Fever
  * Unexplained weight loss
  * Loss of appetite
  * Hemoptysis
  * Shortness of breath
  * Chest pain
  * Night sweats
  * Fatigue
* Suggestive TB on chest x-ray based on pulmonologist or internist consultant of pulmonology opinion
* Age ≥ 18 years' old
* Willing to be treated or evaluated at study site
* Willing to have specimens stored for use in future studies
* Patient denies having TB treatment for more than 7 days in the last 1 month (30 days).

Exclusion Criteria:

Pregnancy or any serious condition includes, but not limited to, liver disease, chronic kidney disease, and psychiatric illness that might interfere with study compliance (based on the clinician judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presumptive TB patients, >=18 years old. This study will analyze 500 subjects bacteriologically confirmed TB (250 new cases and 250 previously treated cases). To obtain the numbers, we estimate to enroll 1357 subjects presumptive TB (1000 new cases and 357 previously treated cases). These numbers are made based on our estimation that 25% of presumptive new TB cases and 70% of presumptive previously treated TB cases will be bacteriologically confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. dr. Erlina Burhan, SpP(K), MSc, Principal Investigator — Persahabatan Hospital, Jakarta
Locations (7):
- Indonesia (7):
  - Site 520: University of Udayana/Sanglah Hospital, Denpasar, Bali
  - Site 560: University of Diponegoro/ Dr. Kariadi Hospital, Semarang, Central of Java
  - Site 590: Persahabatan Hospital, Jakarta, DKI Jakarta
  - Site 570: University of Airlangga/ Dr. Soetomo Hospital, Surabaya, East of Java
  - Site 600 : Adam Malik Hospital, Medan, North Sumatra
  - Site 550: University of Hassanudin/ Dr. Wahidin Sudirohusodo Hospital, Makassar
  - Site 580: University of Gadjah Mada/ Dr. Sardjito Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February 2017 through November 2018. The study was done at 7 hospitals in Indonesia.
Pre-assignment Details: From total target 1357 subjects, only achieved 490 subjects enrolled.
Groups:
- Presumptive TB: TB patients with cough for 2 weeks or longer with at least one additional TB symptom and a chest x-ray suggestive of TB.
Period: Overall Study
Arm/Group | Presumptive TB
Started | 490
Completed | 447
Not Completed | 43
Not completed — Investigator discretion | 43

BASELINE CHARACTERISTICS:
Population: TB patients with cough for 2 weeks or longer with at least one additional TB symptom and a chest x-ray suggestive of TB.
Arm/Group | Presumptive TB
Number analyzed (Participants) | 447
Age, Categorical [Count of Participants; unit: Participants] — Population: Total excluded was 43 participants
  Participants
    <=18 years | 0
    Between 18 and 65 years | 426
    >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total excluded was 43 participants
  Participants
    Female | 173
    Male | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total excluded was 43 participants
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 447
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total excluded was 43 participants
  Participants
    American Indian or Alaska Native | 0
    Asian | 447
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of MDR TB Cases Amongst New TB Cases and Previously Treated TB Cases
Description: AFB smear and GeneXpert were performed at the microbiology laboratory of the study site. Culture and drug susceptibility tests were conducted at appointed National TB Program Reference Laboratories.
Time Frame: 2 months after enrollment
Population: TB cases with bacteriologically confirmed TB with positive MTB culture
Measure: Count of Participants; unit: Participants
Groups:
- MDR TB Amongst New TB Cases: New TB cases with bacteriologically confirmed TB with positive MTB culture and categorized as having MDR-TB
- MDR TB Amongst Previously Treated TB Cases: Previously treated TB cases with bacteriologically confirmed TB with positive MTB culture and categorized as having MDR-TB
Arm/Group | MDR TB Amongst New TB Cases | MDR TB Amongst Previously Treated TB Cases
Number analyzed (Participants) | 260 | 187
Participants | 23 | 64

2. Secondary Outcome: Number of Participants Who Were Cured, Failed, Died, Treatment Completion, and Lost to Follow-up
Description: From 447 subjects with all sputum examination results, only 328 subjects confirmed by bacteriology and the treatment outcome were categorized as followed:
  1. Cured
  2. Failed
  3. Died
  4. Treatment completion
  5. Lost to follow up
Time Frame: 12- 30 months
Population: The proportion of treatment outcomes from all subjects with bacteriologically confirmed (n=328 subjects)
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Outcome: The proportion of treatment outcomes from all subjects with bacteriologically confirmed (n=328 subjects)
Arm/Group | Treatment Outcome
Number analyzed (Participants) | 328
Participants
  Cured | 222
  Failed | 12
  Died | 31
  Treatment complete | 15
  Treatment lost to follow-up | 48

3. Secondary Outcome: Factors for Treatment Success.
Description: Protective factors were collected by interview with the subjects. 237 subjects with confirmed bacteriologically and cured or complete treatment were analyzed for this outcome.
Time Frame: 12-30 months
Population: Treatment success was defined as cured or complete treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Success Factors: Treatment success was defined as cured or complete treatment.
Arm/Group | Treatment Success Factors
Number analyzed (Participants) | 237
Participants
  Males | 143
  Non-Smoking Group | 204
  Normal/overweight (BMI>=18) | 125
  New TB cases | 146
  Lung lesion in CXR > 2 zones | 175

4. Secondary Outcome: Factors of Treatment Interruption.
Description: Risk factors of treatment interruption were collected by interview with the subject. 91 subjects were defined as lost to follow-up or treatment failure or died and analyzed for this outcome.
Time Frame: 12-30 months
Population: Risk factors of treatment interruption were collected by interview with the subject. 91 subjects were defined as lost to follow-up or treatment failure or died and analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Interruption: Treatment interruption was defined as lost to follow-up or treatment failure or died.
Arm/Group | Treatment Interruption
Number analyzed (Participants) | 91
Participants
  Male group | 56
  Non-smoking group | 81
  Underweight (BMI<18) | 51
  Previously treated | 54
  Lung lesion in CXR >2 zones | 75

5. Secondary Outcome: TB Case Category
Description: TB category was defined as clinically TB or bacteriologically confirmed TB. 447 subjects with sputum examination were analyzed for this outcome.
Time Frame: 12-30 months
Population: TB category was defined as clinically TB or bacteriologically confirmed TB. 447 subjects with sputum examination were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Clinically TB: Clinically TB was defined when the subjects have cough >= 2 weeks, have at least 1 other TB symptoms and suggestive TB on chest X-ray and none of the laboratory results were positive.
- Bacteriologically Confirmed TB: Bacteriologically confirmed TB was defined when at least one of the three examinations (AFB, GeneXpert, culture) was positive.
Arm/Group | Clinically TB | Bacteriologically Confirmed TB
Number analyzed (Participants) | 447 | 447
Participants | 99 | 348

6. Secondary Outcome: The Performance of AFB and Xpert MTB/RIF
Description: Assess the sensitivity and specificity of AFB and Xpert MTB/RIF to culture as gold standard.
  312 subjects had positive sputum culture were used for evaluation of sensitivity. Meanwhile, 99 subjects that had no bacterial evidence of MTB infection (AFB, culture, and Xpert negative) and 36 subjects that were only AFB and/or Xpert MTB/RIF positive were used to evaluate the specificity. In total 135 subjects were analyzed to evaluate the specificity.
Time Frame: 12-30 months
Population: Assess the sensitivity and specificity of AFB and Xpert MTB/RIF to culture as gold standard.
  312 subjects had positive sputum culture were used for evaluation of sensitivity. Meanwhile, 99 subjects that had no bacterial evidence of MTB infection (AFB, culture, and Xpert negative) and 36 subjects that were only AFB and/or Xpert MTB/RIF positive were used to evaluate the specificity. In total 135 subjects were analyzed to evaluate the specificity.
Measure: Count of Participants; unit: Participants
Groups:
- Sensitivity AFB; Sensitivity Xpert MTB/RIF: Subjects that had positive sputum culture were used for evaluation of sensitivity.
- Specificity AFB; Specificity Xpert MTB/RIF: Subjects that had no bacterial evidence of MTB infection (AFB, culture, and Xpert negative) and subjects that were only AFB and/or Xpert MTB/RIF positive were used to evaluate the specificity.
Arm/Group | Sensitivity AFB | Specificity AFB | Sensitivity Xpert MTB/RIF | Specificity Xpert MTB/RIF
Number analyzed (Participants) | 312 | 135 | 312 | 135
Participants | 269 | 117 | 304 | 99

7. Secondary Outcome: The Performance of Xpert MTB/RIF
Description: Assess the performance of Rifampicin susceptibility results in Xpert MTB/RIF against result in drug susceptible test (DST) as gold standard.
  312 subjects had positive sputum culture were used to assess the performance of Xpert MTB/RIF.
  196 subjects were sensitive to Rif in Xpert MTB/RIF. While 116 subjects had resistant to Rif in Xpert MTB/RIF.
Time Frame: 12-30 months
Population: Assess the performance of Rifampicin susceptibility results in Xpert MTB/RIF against result in drug susceptible test (DST) as gold standard.
  312 subjects had positive sputum culture were used to assess the performance of Xpert MTB/RIF.
  196 subjects were sensitive to Rif in Xpert MTB/RIF. While 116 subjects had resistant to Rif in Xpert MTB/RIF.
Measure: Count of Participants; unit: Participants
Groups:
- DST Sensitive: Subjects with sensitive to Rif in Xpert MTB/RIF.
- DST Resistant: Subjects with resistant to Rif in Xpert MTB/RIF.
Arm/Group | DST Sensitive | DST Resistant
Number analyzed (Participants) | 196 | 116
Participants
  Xpert negative | 6 | 2
  Xpert sensitive | 165 | 2
  Xpert resistant | 25 | 112

ADVERSE EVENTS:
Time Frame: 12-30 months
Description: any untoward or unfavorable medical occurrence in a human subject that occurs within 48 hours of a study-related blood draw that is possibly, probably, or definitely related to the blood draw. Any event outside of this 48 hour window period will not be considered an AE for this study.
Groups:
- Presumptive TB: Presumptive TB patients
Arm/Group | Presumptive TB
All-Cause Mortality (participants affected / at risk) | 65/447
Serious Adverse Events (participants affected / at risk) | 0/447
Other Adverse Events (participants affected / at risk) | 0/447

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT02758236/Prot_SAP_ICF_000.pdf